CLINICAL TRIAL: NCT00004129
Title: Phase I/II Study of Interstitial Colloidal 32P for the Treatment of Recurrent Malignant Central Nervous System Tumors and Primary Central Nervous System Tumors With Poor Prognostic Factors
Brief Title: Phosphorus 32 in Treating Patients With Glioblastoma Multiforme
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Center for Molecular Medicine (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000067357; CMM-2; NCI-V99-1575
Record Dates: First submitted 1999-12-10; First posted 2003-01-27 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2008-04

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: recurrent adult brain tumor; adult glioblastoma; adult giant cell glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Brain Neoplasms; Glioblastoma; Gliosarcoma | interventions — Brachytherapy; Phosphorus-32

INTERVENTIONS:
Radiation: brachytherapy
Radiation: phosphorus P32

SUMMARY:
RATIONALE: Radioactive drugs such as phosphorus 32 may be able to kill tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of phosphorus 32 in treating patients with glioblastoma multiforme.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the dosimetry toxicity of interstitial colloidal phosphorus P32 (C P32) in patients with recurrent or poor prognosis grade 4 astrocytoma.
* Determine the maximum tolerated dose of C P32 administered directly into the tumor of these patients.
* Determine the maximum tolerated fractionated dose of interstitial C P32 in these patients.
* Determine the therapeutic response rate to the acceptable single and fractionated doses of C P32 in these patients.

OUTLINE: This is a dose-escalation study.

Patients receive interstitial colloidal phosphorus P32 (C P32) on day 0. Courses repeat every 4-6 weeks in the absence of disease progression or unacceptable toxicity.

Cohorts of 3 patients receive escalating doses of C P32 until the maximum tolerated dose (MTD) is determined. The MTD is defined the dose at which 2 of 3 patients experience dose-limiting toxicity.

Patients are followed at 1, 2, 4, 6, 9, 15, and 24 weeks.

PROJECTED ACCRUAL: A minimum of 12 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven grade 4 astrocytoma (glioblastoma)

  * Failed external beam radiotherapy and/or surgery OR
  * Poor prognosis disease
* No clinical evidence of metastatic disease within the CNS other than the primary tumor site
* Stereotactic biopsy or gross total excision with residual tumor
* Lesion 3 to 5 cm in size
* No spinal cord tumor(s)

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 70-100%

Life expectancy:

* Not specified

Hematopoietic:

* WBC at least 3,000/mm3
* Neutrophil count at least 1,900/mm3
* Platelet count at least 100,000/mm3
* Hemoglobin at least 9 g/dL (transfusion allowed)

Hepatic:

* Not specified

Renal:

* Creatinine no greater than 1.5 mg/dL
* BUN less than 25 mg/dL

Other:

* Not pregnant
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Not specified

Endocrine therapy:

* Not specified

Radiotherapy:

* See Disease Characteristics

Surgery:

* See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 1999-09

CONTACTS AND LOCATIONS:
Overall Officials: Stanley E. Order, MD, ScD, FACR, Study Chair — Center for Molecular Medicine
Locations (1):
- Center for Molecular Medicine, Garden City, New York, United States